CLINICAL TRIAL: NCT05018897
Title: Randomized Controlled Trial of a Strategic Disclosure Intervention for Suicide Attempt Survivors
Brief Title: Strategic Disclosure Intervention for Suicide Attempt Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Illinois Institute of Technology (Other)
Collaborators: Depression and Bipolar Support Alliance (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: YIG-1-151-19
Record Dates: First submitted 2021-06-01; First posted 2021-08-24 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Suicide, Attempted; Mood Disorders
Keywords: peer intervention; virtual intervention; suicide; disclosure
MeSH Terms: conditions — Suicide, Attempted; Mood Disorders; Suicide

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two comparison groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- To Share or Not to Share (Experimental): Manualized, peer-led, strategic disclosure program to guide participants in disclosing suicidality, held in group format, consisting of six sessions, each one hour in duration, once per week.
  Pre-survey, post-survey, and 3-month follow-up survey
  Interventions: Behavioral: To Share or Not to Share
- Peer Support (Active Comparator): Peer-led support group, held in group format, consisting of six sessions, each one hour in duration, once per week.
  Pre-survey, post-survey, and 3-month follow-up survey
  Interventions: Behavioral: Peer Support

INTERVENTIONS:
Behavioral: To Share or Not to Share — Strategic disclosure intervention to help participants evaluate the pros and cons of disclosing suicidality and provide guidance on best way to disclose to get needs met. Six one-hour virtual sessions conducted weekly.
  Arms: To Share or Not to Share
Behavioral: Peer Support — Peer-led support group for mood disorders. Six one-hour virtual sessions conducted weekly.
  Arms: Peer Support

SUMMARY:
While suicide prevention depends on people disclosing suicidal thoughts and behaviors in order to get help, those who talk about their suicidality also face negative responses from the people who they tell. The investigators will conduct a randomized controlled trial of a peer-led strategic disclosure intervention for suicide attempt survivors (The To Share or Not to Share Program; called 2Share). This study evaluates the impact of the intervention on suicidal thoughts and behaviors, depression, stigma, disclosure behaviors, and psychosocial outcomes.

DETAILED DESCRIPTION:
The estimated 1.3 million Americans who survive a suicide attempt suicide each year are at risk for ongoing suicide ideation, repeated suicide attempts, and ultimately dying by suicide. While suicide prevention often depends on people openly discussing suicidal thoughts and behaviors in order to get help for themselves or others, those who talk about their suicidality often face negative reactions from confidants. Stigmatizing responses in the form of stereotypes, prejudice, and discrimination may exacerbate symptoms and interfere with social relationships, employment opportunities, and help seeking. Feelings of shame and rejection are common experiences of suicide attempt survivors and the mere anticipation of rejection can encourage attempt survivors to maintain their silence.

Research suggests that suicide disclosure could help suicide attempt survivors in attaining needed care, expanding social support networks, strengthening relationships, and advancing coping strategies. However, few interventions are available to assist suicide attempt survivors in making critical disclosure decisions.

A peer-led strategic disclosure intervention (The 2Share Program), developed through a collaborative process with suicide attempt survivors, aids participants in: (a) evaluating the benefits and risks of disclosure; (b) considering ways to disclose; and (c) developing disclosure scripts. A pilot randomized controlled trial (RCT) with community-dwelling attempt survivors (n=38) found that intervention participants had significantly decreased depression and internalized stigma, and increased self-esteem as compared with the control group. However, this study was small and did not evaluate changes in suicidal thoughts and behaviors, help-seeking, or disclosure outcomes. The methodology was also limited in measuring longer term outcomes.

Given limitations of past research, the investigators propose a randomized controlled trial of the 2Share strategic disclosure program for community-dwelling suicide attempt survivors. The primary goal of this study is to evaluate the impact of the intervention on suicidal thoughts and behaviors and depression. Secondary goals are to examine intervention impact on stigma, disclosure, and psychosocial outcomes. A final goal of the project is to qualitatively examine participant experiences with disclosure over time.

The proposed research addresses the American Foundation for Suicide Prevention priority of determining what interventions are effective and what prevents individuals from engaging in suicidal behavior. The 2Share intervention is the first to address strategic disclosure in suicide attempt survivors, and this study will provide important data about disclosure that can ultimately aid in understanding suicide prevention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* self-reported diagnosis of mood disorder
* At least one lifetime suicide attempt

Exclusion Criteria:

* a self-reported suicide attempt within the last 3 months
* do have concerns about disclosure/ not willing to participate in program
* do not have email address
* do not have technical capability to connect to virtual platform
* cannot speak or read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in suicidality on the 9-item Suicidal Ideation Attributes Scale (SIDAS) at Week 6 and Week 19 | Baseline, Week 6, Week 19
  The SIDAS is a validated, self-reported instrument assessing suicidality over the past month. Possible item scores range from 0 (no thoughts) to 10 (always) Change = (Week 6 Score - Baseline Score), (Week 19 - Baseline Score)
Change from Baseline in depression on the 10- item Center for Epidemiologic Studies Depression Scale (CESD-10) at Week 6 and Week 19 | Baseline, Week 6, Week 19
  he CESD-10 is a validated, self-reported instrument assessing depression over the past week. Possible item scores range from 1 (rarely to none of the time) to 4 (most or all of the time)

SECONDARY OUTCOMES:
Change from Baseline in internalized stigma on the 9- item Internalized Stigma of Suicide (ISSA) at Week 6 and Week 19 | Baseline, Week 6, Week 19
  The ISSA is a validated, self-reported instrument assessing internalized stigma. Possible item scores range from 1 (strongly disagree) to 4 (strongly agree) Change = (Week 6 Score - Baseline Score), (Week 19 - Baseline Score)
Change from Baseline in stigma-related stress on the 8- item Suicide Stigma Stress Scale (4S) at Week 6 and Week 19 | Baseline, Week 6, Week 19
  The 4S is a validated, self-reported instrument assessing stigma-related stress Possible item scores range from 1 (strongly disagree) to 7 (strongly agree) Change = (Week 6 Score - Baseline Score), (Week 19 - Baseline Score)
Change from Baseline in self-esteem on the 10- item Rosenberg Self-Esteem (RSE) scale at Week 6 and Week 19 | Baseline, Week 6, Week 19
  The RSE is a validated, self-reported instrument assessing self-esteem. Possible item scores range from 1 (strongly disagree) to 5 (strongly agree) Change = (Week 6 Score - Baseline Score), (Week 19 - Baseline Score)
Change from Baseline in disclosure self-efficacy on the 2- item Disclosure Self-Efficacy (DSE) scale at Week 6 and Week 19 | Baseline, Week 6, Week 19
  The DSE is a validated, self-reported instrument assessing self-efficacy in disclosing suicidality. Possible item scores range from 1 (not at all) to 7 (very much) Change = (Week 6 Score - Baseline Score), (Week 19 - Baseline Score)
Change from Baseline in secrecy on the 14- item Self-Harm and Suicide Disclosure Scale (SHSDS) at Week 6 and Week 19 | Baseline, Week 6, Week 19
  The SHSDS scale is a validated, self-reported instrument assessing disclosure of suicidality. Items are answered yes/no and focus on disclosure of particular ideations and behaviors.
  Change = (Week 6 Score - Baseline Score), (Week 19 - Baseline Score)
Change from Baseline in secrecy on the 5- item Secrecy scale at Week 6 and Week 19 | Baseline, Week 6, Week 19
  The Secrecy scale is a validated, self-reported instrument assessing secrecy in disclosing suicidality. Possible item scores range from 1 (strongly disagree) to 7 (strongly agree) Change = (Week 6 Score - Baseline Score), (Week 19 - Baseline Score)
Change from Baseline in mental health seeking on the 3- item Mental Health Seeking Intention scale (MHSIS) at Week 6 and Week 19 | Baseline, Week 6, Week 19
  The MHSIS is a validated, self-reported instrument assessing intention to seek help. Possible item scores range from 1 (extremely unlikely) to 7 (extremely likely) Change = (Week 6 Score - Baseline Score), (Week 19 - Baseline Score)
Change from Baseline in quality of life on the 1- item quality of life scale at Week 6 and Week 19 | Baseline, Week 6, Week 19
  The question asks participants to rate their quality of life. Possible scores range from 1 (very poor) to 5 (very good) Change = (Week 6 Score - Baseline Score), (Week 19 - Baseline Score)
Change from Baseline in social support on the 8- item social support scale at Week 6 and Week 19 | Baseline, Week 6, Week 19
  The Social Support scale is the emotional subscale from the NIH Toolbox for Social Relationships and is a validated, self-reported instrument assessing social support. Possible item scores range from 1 (never) to 5 (always) Change = (Week 6 Score - Baseline Score), (Week 19 - Baseline Score) Change = (Week 6 Score - Baseline Score), (Week 19 - Baseline Score)

CONTACTS AND LOCATIONS:
Locations (1):
- Illinois Institute of Technology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Results will be available through the National Institute of Mental Health (NIMH) Data Archive and through the project website at the National Consortium on Stigma and Empowerment (NCSE). No identifying information will be connected to the data and we do not believe that there is a possibility of deductive disclosure of subjects with unusual characteristics. We will certify the quality of all data prior to submission to New Drugs and Clinical Trials (NDCT). Descriptive/raw data will be submitted semi-annually (prior to January 15 and July 15) and will be checked for quality within four months. All other data will be submitted at the time of publication, or prior to the end of the grant, whichever occurs first. The final de-identified dataset and codebook will be posted on NCSE website at the time of publication. We will share results, positive and negative, specific to the cohorts and outcome measures studied by using the Study functionality.
Time Frame: The final de-identified dataset and codebook will be shared at the time of publication.